CLINICAL TRIAL: NCT01215266
Title: Prospektiv, Randomisierte, Doppelblinde, Multizentrische Phase-II- Studie Zum Vergleich Der Wirksamkeit Einer Chemotherapie Mit Gemcitabin Plus Cisplatin Und Sorafenib (BAY 43-9006) Versus Gemcitabin Plus Cisplatin Und Plazebo in Der Therapie Des Lokal Fortgeschrittenen Bzw. Metastasierten Urothelkarzinoms AB 31/05 - RUTT 204 - SUSE
Brief Title: Sorafenib in Urothelium Cancer of Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Association of Urologic Oncology (AUO) (Other)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AB 31/05 RUTT 204; 2005-006098-29 (EudraCT Number)
Record Dates: First submitted 2010-10-01; First posted 2010-10-06 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Chemotherapy; Urothelium cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib — Day 3-21 2x2 800 mg(milligram) daily
  Other Names: Prüfsubstanz
  Arms: Sorafenib
Drug: Placebo — Day 3-21 2x2 800 mg(milligram) daily
  Other Names: Plazebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the use of Sorafenib additionally to gemcitabine and cisplatin in bladder cancer.

DETAILED DESCRIPTION:
A controlled, double-blind, randomized study to evaluate the influence of Sorafenib in bladder cancer patients additionally to chemotherapy with gemcitabine and cisplatin compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Men and Women > 18 years

* Condition ECOG(Eastern Cooperative Oncology Group) 0-1
* Life expectancy at least 12 weeks
* Women in conceptional age: negative pregnancy test and adequate contraception (oral contraceptive, spiral); at men adequate contraception of the man (condom use) to 3 months after discontinuation of therapy with sorafenib
* Histologically or cytologically proven urothelial carcinoma of the bladder or upper urinary tract
* Locally advanced or metastatic urothelial carcinoma of the bladder or upper urinary tract (T3b,T4/ N+/M+)
* At least one unidimensional measurable lesion on CT(Computed Tomography) or MRI(Magnetic resonance imaging) according to RECIST(Response Evaluation Criteria in Solid Tumors) criteria
* Adequate hematologic, renal, hepatic and coagulation-physiological functions
* Leukocytes > 1.500 cells /ml (per milliliter)
* Hemoglobin >9g/dl(gram per deciliter)
* Platelet > 100000 /ml
* Serum creatinine < 2 x upper limit of normal or creatinine clearance ≥ 45 ml/min (milliliter per minute)
* Total Bilirubin < 1,5 x upper limit of normal
* GOT/GPT (glutamate-oxalacetate-transaminase/glutamate-pyruvate-transaminase) < 2,5 x upper limit of normal, at liver metastases < 5x upper limit of normal
* alkaline phosphates < 5 x upper limit of normal
* Amylase/ Lipase < 1,5 x upper limit of normal
* INR(International Normalized Ratio) und PTT(Partial Thromboplastin Time) < 1,5 x upper limit of normal
* Informing the patient about the study and the present written consent to participate after clarification in accordance with the stipulations of AMG(german drug law), and the principles of the Ethics Committee ("informed consent").

Exclusion Criteria:

* Absence of the above inclusion criteria
* Dialysis after nephrectomy
* Patients with brain tumors and / or brain metastases
* Previous or existing serious cardiovascular (grade III - IV according to NYHA(New York Heart Association)) disease, active angina pectoris or ischemia, myocardial infarction within 6 months prior to enrollment, or patients with serious cardiac arrhythmias requiring antiarrhythmic therapy (beta blockers and digoxin are permitted)
* Patients with uncontrolled high blood pressure, systolic blood pressure> 150 mm Hg or diastolic pressure> 90 mmHg despite optimal medical treatment
* Patients with thrombotic or embolic events such as stroke or pulmonary embolism
* Patients with recently or known bleeding diathesis
* Known significant neurological or psychiatric diseases including dementia and epileptic seizures
* Serious inflammatory eye disease, hearing impairment
* Pulmonary (pO2(Blood oxygen) <60 mm Hg(Millimeters of mercury)), hematopoietic (eg(exempli gratia) severe bone marrow aplasia), hepatic or renal disease
* Patients with poorly controlled diabetes mellitus
* Serious bacterial or fungal infections(>Grade 2 NCI-CTC(National Cancer Institute-Common Terminology Criteria) Version 3)
* chronic hepatitis B or C, HIV(human immunodeficiency virus) infection
* Autoimmune disease
* Allergic reactions to be used in respect of a drug
* prior organ transplantation
* prior autologous bone marrow transplant or stem cell transferred within the last 4 months before study
* Manifesto, second malignancy or other malignancy within the past 5 years (except basal cell carcinoma, carcinoma in situ of the cervix, incidental prostate carcinoma)
* Pregnancy or breast-feeding
* Lack of cooperation and the ability to cooperate, predictable problems with the aftercare, psychiatric disorders, substance abuse, lack of capacity of the patient
* Participation in other treatment studies in the last 4 weeks
* Previous treatment with chemotherapy or immunotherapy
* Simultaneous treatment with other anti-tumor therapies after study start
* Intravesical chemotherapy within the last 4 weeks
* Irradiation within the last 4 weeks
* Previous radiation therapy, when all were irradiated to the assessment of tumor response used lesions
* Complex operations, open biopsy or significant injuries within the last 4 weeks before study
* Serious wound healing disorder, ulcers or bone fractures in the last 4 weeks before study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 5 years

SECONDARY OUTCOMES:
Response rates, time of response | 5 years
Time to progression | 5 years
Overall survival | 5 years
Evaluation and comparison in both treatment arms | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Krege, Prof. Dr., Study Chair — Universität Duisburg-Essen